CLINICAL TRIAL: NCT03020628
Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess the Immunogenicity and Safety of 'NBP607-QIV(Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine)' in Children Aged 6~35 Months
Brief Title: Immunogenicity and Safety of Quadrivalent Influenza Vaccine in Children Aged 6~35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607-QIV_FluC_III_2016
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Influenza, Human
Keywords: Influenza Vaccines; Vaccines, Inactivated; Cell Culture-Derived
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NBP607-QIV 0.5mL (Experimental): Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine
  Interventions: Biological: NBP607-QIV
- NBP607-TIV 0.25mL (Active Comparator): Trivalent Inactivated Cell Culture-derived Influenza Vaccine
  Interventions: Biological: NBP607-TIV

INTERVENTIONS:
Biological: NBP607-QIV — For subjects 6 months to 35 months of age, Single dose administration, Intra-muscular [* 2 doses for subjects without influenza vaccination history, administered at least 4 weeks apart]
  Arms: NBP607-QIV 0.5mL
Biological: NBP607-TIV — For subjects 6 months to 35 months of age, Single dose administration, Intra-muscular [* 2 doses for subjects without influenza vaccination history, administered at least 4 weeks apart]
  Arms: NBP607-TIV 0.25mL

SUMMARY:
This study is a multi-center, randomized, double-blind Phase III Clinical trial. The purpose of this study is to assess the immunogenicity and safety of the quadrivalent cell culture-derived influenza vaccine compare to the trivalent cell culture-derived influenza vaccine in children aged 6~35 months.

DETAILED DESCRIPTION:
Subjects are randomly assigned in a 2:1 ratio to NBP607-QIV 0.5mL versus NBP607-TIV 0.25mL. To assess the immunogenicity, antibody levels are evaluated by hemagglutination inhibition(HI) assay from sera obtained at pre-vaccination and 28 days post-vaccination. To assess the safety, solicited adverse events for 7 days post-vaccination and unsolicited adverse events for 28 days post-vaccination are assessed and reported. The serious adverse events are collected during 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 35 months
* Those who was born after normal pregnancy period(37 weeks) for aged 6 months to < 1 year
* Those whose legally acceptable representative have given written consent to participate in the study and comply with all study requirements.

Exclusion Criteria:

* Subjects with immune deficiency disorder or malignant cancer.
* History of any hypersensitivity following administration of vaccine or Guillain-Barre syndrome.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subjects who experienced fever within 72 hours before vaccination or with the febrile disease(exceeding 38.0℃) on screening day.
* Subjects who had received immunosuppressant or immune-modifying drug within 3 months before screening.
* Subjects who had received blood products or immunoglobulin within 3 months before screening.
* Subjects who had received influenza vaccination within 6 months prior to the screening.
* Subjects who had received other vaccination within a month before screening, or those who had another vaccination scheduled within a month after study vaccination.
* Subjects who had received any other investigational products within 4 weeks prior to study vaccination.
* Subjects with clinically significant chronic disease.
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
HI[hemagglutination Inhibition] derived parameters: Seroprotection rate(a lower bound of 95% CI) > 70% | At Day 28 post-vaccination
  Seroprotection rate is the proportion of subjects achieving a post-vaccination HI titer ≥ 1:40
HI[hemagglutination Inhibition] derived parameters: Seroconversion rate(a lower bound of 95% CI) > 40% | At Day 28 post-vaccination
  Seroconversion is defined as a pre-vaccination HI titer of <1:10 with a post-vaccination titer ≥ 1:40, and a significant increase was defined as at least a four fold increase in HI titer
HI[hemagglutination Inhibition] derived parameters: GMR (a lower bound of 95% CI) > 2.5 | At Day 28 post-vaccination
  GMR [geometric mean ratio, mean fold increase]

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kyung Kim, Study Chair — Korea University Ansan Hospital; Hye Kyung Cho, Principal Investigator — Gachon University Gil Medical Center; Ki Hwan Kim, Principal Investigator — Incheon St.Mary's Hospital; Byung Wook Eun, Principal Investigator — Eulji General Hospital; Yae Jean Kim, Principal Investigator — Samsung Medical Center; Jina Lee, Principal Investigator — Asan Medical Center; Dong Ho Kim, Principal Investigator — Korea Institute of Radiological and Medical Science; Hwang Min Kim, Principal Investigator — Wonju Severance Christian Hospital; Nam Hee Kim, Principal Investigator — Inje University Ilsan Paik Hospital; Dae Sun Jo, Principal Investigator — Chonbuk National University Hospital; Eun Young Cho, Principal Investigator — Chungnam National University Hospital; Seon Hee Shin, Principal Investigator — Hallym University Dongtan Sacred Heart Hospital
Locations (12):
- South Korea (12):
  - Korea University ANSAN hospital, Ansan
  - Chungnam National University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - Gachon University Gil Medical center, Incheon
  - The Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Asan Medical Center, Seoul
  - Eulji General Hospital, Seoul
  - Hallym University Dongtan Sacred Heart Hospital, Seoul
  - Korea Institute of Radiological and Medical Science, Seoul
  - Samsung Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No